CLINICAL TRIAL: NCT01542021
Title: Establishing a Neo-Adjuvant Platform for Developing Targeted Agents: Androgen Deprivation Therapy Prior to Prostatectomy for Patients with Intermediate and High Risk Prostate Cancer
Brief Title: Androgen Deprivation Therapy Prior to Prostatectomy for Patients with Intermediate and High Risk Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-182
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Prostatic Adenocarcinoma
Keywords: prostate; Degarelix; injections; radical prostatectomy; 11-182
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Untreated patients degarelix injection occur at days 4± 1 (Experimental): Treatment will consist of a single 240 mg injection of degarelix 4 ± 1 day before radical prostatectomy
  Interventions: Drug: degarelix injection
- Untreated patients degarelix injection occur at days and 7± 1. (Experimental): Treatment will consist of a single 240 mg injection of degarelix 7±1 day before radical prostatectomy
  Interventions: Drug: degarelix injection
- treated patients with androgen deprivation (Experimental): Patients already treated with androgen deprivation are assigned to Cohort 3 and maintained on current androgen deprivation therapy until they undergo or have already undergone RP at MSKCC. Will include patients who have already undergone hormonal therapy (of any duration between 1 and 6 months) prior to prostatectomy.
  Interventions: Drug: androgen deprivation therapy
- Untreated patients degarelix injection occur at days 14±1 (Experimental): Treatment will consist of a single 240 mg injection of degarelix 14±1 day before radical prostatectomy
  Interventions: Drug: degarelix injection

INTERVENTIONS:
Drug: degarelix injection — Treatment will consist of a single 240 mg injection of degarelix 4 ± 1 day before radical prostatectomy, depending on treatment arm.
  Arms: Untreated patients degarelix injection occur at days 4± 1
Drug: degarelix injection — Treatment will consist of a single 240 mg injection of degarelix 7 ± 1 day before radical prostatectomy, depending on treatment arm.
  Arms: Untreated patients degarelix injection occur at days 14±1; Untreated patients degarelix injection occur at days and 7± 1.
Drug: androgen deprivation therapy
  Arms: treated patients with androgen deprivation

SUMMARY:
Degarelix is an approved drug that is used to treat prostate cancer by lowering testosterone levels in the body.

Degarelix is commonly given with radiation for prostate cancer, but less frequently with surgery since there has been no proven benefit with this approach.

The investigators do not expect the patient to benefit directly from treatment with degarelix since their prostate will be removed shortly after the drug is given. Instead, the investigators hope to learn about how degarelix and other treatment that lowers your testosterone effects prostate cancer cells and use this information to develop better treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of prostatic adenocarcinoma by MSKCC inclusive of the following:
* 3 or more positive biopsy cores or equivalent tumor specimen as confirmed by pathologist
* At least 2 cores containing ≥3 mm of tissue with carcinoma or equivalent tumor specimen as confirmed by pathologist
* A primary tumor Gleason score ≥ 7
* Adequate primary biopsy tissue or equivalent tumor specimen as confirmed by pathologist available for protocol required analysis (i.e. bladder or TURP specimen)
* Planning to have or have had a radical prostatectomy (RP) at MSKCC
* Candidates may have a history of deep vein thrombosis, pulmonary embolism, and/or cerebrovascular accident, or require concomitant systemic anticoagulation, if otherwise deemed to be suitable for RP
* Karnofsky performance status >70% (Appendix A)
* Sexually active fertile subjects, and their partners, must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 3 months after the dose of study drug(s) for Cohorts 1 , 2 and 4, and for 3 months after the surgery for Cohort 3
* For cohorts 1,2 and 4 only:, non-castrate testosterone level (>100 ng/dL)
* For cohort 3 only:, 1-6 months of androgen deprivation therapy (gonadotropin hormone releasing analogs with or without an anti-androgen) prior to prostatectomy with a castrate testosterone level of <50 ng/dL within 1 month prior to prostatectomy.

Exclusion Criteria:

* Histologic variants in the primary tumor (histologic variants other than adenocarcinoma)
* Current or prior chemotherapy
* The use of the 5-alpha-reductase inhibitor dutasteride must be discontinued within 4 weeks of degarelix injection for Cohort 1, 2 and 4, and within 4 weeks of surgery for Cohort 3.
* Saw palmetto administered with the intent to treat the patient's malignancy within 1 week of degarelix injection for Cohorts 1, 2 and 4, and for within 1 week of surgery for Cohort 3
* Current or prior radiation therapy to the prostate
* Active infection or intercurrent illness
* Concomitant therapy with any other experimental drug
* For cohorts 1, 2 and 4 only:, current or prior hormonal therapy (e.g., gonadotropin hormone releasing analogs, megestrol acetate, or antiandrogens) are exclusionary

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-02-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
To assess between the time to determine the time of the maximal change in prostate cancer cell proliferation (Ki-67) and apoptosis rates (cleaved caspase-3) | 2 years
  The primary endpoint is the change in the rate of proliferation (Ki-67) and the rate of apoptosis (cleaved caspase-3), as evaluated by IHC in anatomically matched tumor foci from the pre-treatment diagnostic biopsy and the RP specimen. The levels in pre-treatment biopsy serve as the baseline. Ki-67 is a widely accepted nuclear marker for cell proliferation. Cleaved caspase-3 has been shown to be a reliable marker of apoptosis and correlate with results from other apoptosis markers such as cleaved PARP-1 and TUNEL assay.

SECONDARY OUTCOMES:
To explore the association between PTEN status and maximal changes in prostate cancer proliferation and apoptosis rates in patients treated with androgen deprivation therapy | 2 years
  The secondary endpoint is PTEN status by IHC in the diagnostic biopsy and RP specimens. PTEN status will be determined by an IHC method that has been validated using control prostate cell lines and tissues at MSKCC. The PTEN status will be reported in binary fashion as "retained" (diffuse moderate immunoreactivity retained in benign glands as well as adenocarcinoma on 100X magnification) or "null" (complete loss of nuclear and cytoplasmic immunoreactivity in tumor cells while expression is retained in surrounding stroma.
To explore the association between PI3K pathway (pAKT and pS6) and prostate cancer proliferation and apoptosis rates after treatment with androgen deprivation therapy in relation to other markers of prostate cancer (ERG, AR and NCOA2). | 2 years
  Additional exploratory endpoints include IHC staining for markers of PI3K pathway (pAKT and pS6) as well as other markers of prostate cancer (ERG, AR and NCOA2) in the diagnostic biopsy and RP specimens. Some of these markers have been validated at MSKCC (pS6, ERG), while others (AR, pAKT, NCOA2) are currently being validated and standardized for the study using appropriate cell line and tissue controls. A general semiquantitative scoring method will be used for these markers.
To discover novel biomarkers and correlates of response | 2 years
  through expression profiling of prostate cancer after three time intervals of androgen deprivation therapy and correlate with PTEN and ERG status, proliferation rate, apoptotic rate, and histologic response

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/